CLINICAL TRIAL: NCT03569358
Title: Safety, Tolerability, and Early Efficacy of Immersive Virtual Reality for Early Neurocognitive Stimulation in the Intensive Care Unit.
Brief Title: Immersive Virtual Reality in Mechanically Ventilated Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changi General Hospital (Other)
Collaborators: BetaSight Technologies Pte Ltd (Unknown); Institute for Infocomm Research (Other)
Responsible Party: Principal Investigator, Jessica Quah Li Shan, Associate Consultant, Changi General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 201802-00023
Record Dates: First submitted 2018-05-22; First posted 2018-06-26 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Mechanical Ventilation; Virtual Reality; Delirium
Keywords: Randomised Controlled Study; Unblinded; Electroencephalogram; Feasibility
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual Reality and EEG Interventions (Experimental): In the interventional arm, 20 subjects will receive twice daily sessions of immersive virtual reality for a maximum of 15 minutes, with EEG headband recording starting 5 minutes prior to and 5 minutes after the intervention, for a maximum of 4 consecutive days.
  Interventions: Device: Immersive Virtual Reality; Device: EEG headband
- EEG Intervention group (Active Comparator): In the control arm, 10 subjects would have EEG recorded for 25 mins twice daily, with a minimum of 4 hours intervening, for 3 consecutive days, with the EEG headband. There would be no immersive virtual reality sessions.
  Interventions: Device: EEG headband
- Healthy Volunteers (Active Comparator): At the completion of the above intensive care study recruitment, demographic data of the interventional immersive virtual reality arm would analysed to recuit 10 age-matched healthy volunteers with no known cognitive disorders or visual impairment. This is to compare study data with healthy controls. A 25 minute session consisting of 15 minutes of immersive virtual reality and 5 minutes of EEG recording with the EEG headband before and after the intervention would be performed. Eye-tracking and EEG data from these groups of patients would be compared against subjects in both arms of the study performed in the intensive care unit to investigate for exploratory differences.
  Interventions: Device: Immersive Virtual Reality; Device: EEG headband

INTERVENTIONS:
Device: Immersive Virtual Reality — The immersive virtual reality headgear used is the commercially available FOVE VR headset. It incorporates a 2560x1440 pixel display, position tracking-and eye-tracking. The headset weight 520g with adjustable velcro straps. Softwares are run via a computer connected by HDMI or USB cables.
  Arms: Healthy Volunteers; Virtual Reality and EEG Interventions
Device: EEG headband — The EEG headband is commercially available MUSE band. It incorporates 4-channel dry electrode EEG system where data can be recorded with bluetooth connection.

SUMMARY:
New or worsening cognitive impairment occurs in up to 58% of survivors of critical illnesses and are long-lasting with significant disability and socioeconomic cost. There are currently no known interventions that reduce the incidence of cognitive impairment after critical illnesses. Immersive Virtual Reality (IVR) is the use of technology to create a perception of presence in a three-dimensional, computer-generated interactive simulated environment. Prior clinical studies have demonstrated potential efficacy in rehabilitation of severe traumatic brain injury.

The investigators propose a preliminary study for the evaluation of safety, tolerability, and early efficacy of immersive virtual reality for early neurocognitive stimulation in critically-ill, mechanically ventilated patients. The investigators hypothesize that the use of IVR technology for early neurocognitive simulation is safe and tolerable in these patients. This study will also evaluate whether early application of IVR in critically ill, mechanically ventilated subjects, can provide neurocognitive stimulation.

30 patients admitted to the intensive care unit for acute respiratory failure or septic shock will be evaluated for recruitment. 10 patients will be in the control group and 20 patients would have 2 sessions of IVR planned daily for a maximum of 3 days. Assessment of safety will involve monitoring for physiological derangements in heart rate, respiratory rate, pulse oximetry and blood pressure during the IVR session. Assessment of tolerability will involve monitoring for increased agitation. Assessment of early efficacy will involve evaluation of visual attention during the IVR session. 5-channel electroencephalogram would aim to detect objective changes in visual event-related potentials and the IVR headgear will incorporate eye-tracking technology.

To conclude, should IVR be feasible and safe, future interventional studies may be planned to investigate its impact on reduction in the use of sedatives, analgesia, delirium incidence and severity of cognitive impairment associated with critical illness.

DETAILED DESCRIPTION:
Advancements in the last 2 decades in the field of critical care medicine has led to an improvement in mortality of critically ill patients. This has led to interest in the long-term functional disabilities that the survivors suffer. The risks of developing cognitive dysfunction after critical illness has been associated with older age, longer duration of critical illness, hyperglycaemia, prolonged use of sedatives and analgesia, as well as delirium. The BRAIN-ICU study reported that in adults with respiratory failure and shock, the incidence of cognitive impairment at 1 year was 34% for 1.5 SD below population mean (similar to moderate traumatic brain injury) and 24% for 2.5 SD below population mean (similar to mild Alzheimer's disease). Some proposed mechanisms include cerebral hypoxia secondary to respiratory failure, cerebral inflammation and neuronal apoptosis related to sepsis, and prolonged disruption of sleep cycles. Neuronal imaging such as diffusion-tensor MRI during critical illness show diffuse hyperintense white matter changes and subsequent distant imaging studies show generalised cerebral atrophy.

Critical care societies have endorsed the use of care bundles for pain, agitation and delirium management. Few specialised centres with dedicated survivor clinics evaluate functional impairment via diagnostic investigations, physical, neurological examinations and psychological assessments, to provide personalised rehabilitation. While these initiatives have been shown to improve patient satisfaction, quality of transitional care and reduction of inappropriate emergency room visits, there are no definitive interventions that have improved cognitive outcomes.

Psychiatric co-morbidities of anxiety, depression and post-traumatic stress disorder(PTSD) have been shown to be associated with delirium and cognitive impairment after critical illness. Survivor accounts revealed a mixture of delusional and factual memories resulting in the distortion of experiences. Intensive care diaries involve the recording of significant daily events and is an attempt at systematic reconstruction of memories by medical staff, family and friends. This has been shown to reduce the incidence of PTSD after critical illness. It raises the possibility that incidence of cognitive impairment, too, may be reduced with non-pharmacological methods.

An intensive care admission involves the immersion of a patient in a foreign environment that is dominated by machines, the use of esoteric language by medical staff and persistent sleep disruption that combines deprivation of meaningful sensory stimulation with noxious sensory overload of alarms and lights. There is an unmet need for the provision of a calm, familiar environment, and deliberate neurocognitive simulation with the intention of allowing processes of thought, reasoning, memory and imagination to occur as they do in everyday life. Allowing these cognitive processes to occur may reduce the use of sedatives, delirium occurrence, and possibly cognitive impairment. Cognitive impairment after critical illness is known to decrease the rehabilitation potential of survivors, increase caregiver burden and is associated with higher utilisation of long-term healthcare resources. There is a need for interventional clinical studies that address prolonged cognitive impairment after critical illnesses.

The overall aim of the study is to improve clinical outcomes in critically ill and mechanically ventilated patients.

The primary hypothesis is that the use of an immersive virtual reality headset for early neurocognitive stimulation in critically ill, mechanically ventilated patients is safe and well tolerated (i.e., does not result in significantly increased agitation).

The primary outcome of the study would be the composite endpoint of both safety and tolerability. The immersive VA is considered as safe and tolerable if the patient does not experience any safety or tolerability events. In both arms, subjects who complete of 4 out of 4 to 6 planned sessions would be considered as having met criteria for both safety and tolerability. If 3 or less sessions were initiated, completion of 2 or more sessions would be considered for having met criteria for both safety and tolerability. The IVR intervention would be considered safe and tolerable if the difference in composite endpoint in the intervention arm is not 20% more than the control arm.

Demonstration of safety, defined as the non-occurrence of significant physiological events that require early termination of the IVR session. The use of an iVR is safe and does not cause physiological changes that require the termination of more than 2 out of 6 planned interventions.

Demonstration of tolerability, defined as: the occurrence of the event that the Richmond Agitation-Sedation Score (RASS) greater than or equal to +2 during the use of the immersive virtual reality headset and for the immediate 15 minutes after completion. The RASS score, ranging from -5 to +4, is a validated scoring system used by clinical staff to evaluate the degree of sedation and agitation of mechanically ventilated patients. A score of +2 reflects an agitated state that is characterised by frequent non-purposeful movement or presence of patient-ventilator dys-synchrony. Each subject has 6 planned interventions, completion of 4 out of 6 interventions would be considered demonstration of tolerability.

There are 2 secondary aims in this study to demonstrate early efficacy in terms of neurocognitive stimulation. One would be comparing change in the EEG data after the immersive VR sessions from the baseline, that may indicate visual attention. The hypothesis is that visual attention during the intervention can be demonstrated with EEG waveforms. The other secondary aim will be evaluation of the eye-tracking software as a potential tool for meaningful interaction.

ELIGIBILITY:
Inclusion Criteria:

* Patient Group

  1. Patients aged 21 to 75
  2. Both genders and all races
  3. Acute respiratory failure or septic shock as indications for critical care admission
  4. Anticipated to require mechanical ventilation for a minimum of 48 hours after enrolment
  5. GCS of E3VTM4 or more

Healthy Volunteer Group

1) Age-matched to the subjects of the interventional arm of the ICU subjects.

Exclusion Criteria:

Patient Group

1. Patients who are actively using an interactive device in the intensive care unit prior to enrolment
2. Illnesses with a terminal prognosis within 3 months
3. Prisoners and pregnant patients
4. Blind or deaf patients
5. Premorbid baseline cognitive impairment
6. Neurological diseases affecting cognition as the cause of intensive care admission including but not limited to ischaemic and haemorrhagic strokes, meningitis, encephalitis, traumatic brain injuries and status epilepticus.
7. Severe critical illness with imminent mortality
8. Critical illness requiring the use of paralytic agents
9. Use of vasopressor dose more than an equivalent of Noradrenaline 0.5 mcg/kg/min
10. Use of fractional inspired oxygen on mechanical ventilation of more than 0.8.
11. Presence of external facial, skull vault or cervical injuries, or deformities, precluding the safe application of the VR headset and EEG band.
12. Participation declined by attending intensivist.

Healthy Volunteer Group

1. Known prior neurological or neurocognitive disease.
2. Baseline heart rate more than 100 beats per minute
3. Baseline systolic blood pressure less than 100 mmHg or more than 160 mmHg
4. Respiratory failure requiring supplemental oxygen

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-07-02 (Actual); Primary Completion 2019-07-02 (Estimated); Study Completion 2019-07-02 (Estimated)

PRIMARY OUTCOMES:
The primary outcome of the study would be the number of patients who are able to complete immersive virtual reality session meeting both safety and tolerability criteria. | 4 days
  The IVR intervention would be considered safe and tolerable if the difference in number of subjects having a composite endpoint of both safety and tolerability end-points in the intervention arm is not 20% more than the control arm. Demonstration of safety is the composite of non-occurrence of any 4 physiological events as follows: greater than 30% variability in the heart rate; greater than 30% variability in respiratory rate; systolic blood pressure of less than 90mmHg or more than 160mmHg; pulse oximetry of less than 90%. Demonstration of tolerability is the non-occurrence of the event that Richmond Agitation-Sedation Score (RASS) greater than or equal to +2 during the intervention, sustained for more than 3 minutes.

SECONDARY OUTCOMES:
Exploratory use of EEG changes to quantify differences in attention in delirious mechanically ventilated patients. | 4 days
  EEG data before, during and after the immersive VR sessions would be recorded and compared to subjects in the control arm and the healthy subjects group. The EEG patterns would be translated into an attention score developed by academic collaborator. The hypothesis is that visual and auditory attention during the immersive virtual reality intervention can be demonstrated with EEG signals with differences in the level of attention between subjects who have delirium as assessed by ICU-CAM scores, and those who do not have delirium. The degree of eye blinking and motion artefacts generated during the intervention may also be accurately quantified and compared between intervention and control groups.
Assessment of visual attention in delirious subjects using virtual-reality integrated eye-tracking software. | 4 days
  Assessment of eye movements is a potential tool for assessment of meaningful interaction in mechanically ventilated patients. The subjects would have eye movements recorded during the immersive virtual reality interventions. These would allow identification and quantification of the presence of saccadic eye movements, velocity and duration, as well as the presence and duration of smooth pursuit, to be compared between delirious and non-delirious subjects in the interventional groups.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica LS Quah, M.B.B.S., Principal Investigator — Changi General Hospital
Locations (1):
- Changi General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zimmerman JE, Kramer AA, Knaus WA. Changes in hospital mortality for United States intensive care unit admissions from 1988 to 2012. Crit Care. 2013 Apr 27;17(2):R81. doi: 10.1186/cc12695. PMID 23622086
- [Background] Kaukonen KM, Bailey M, Suzuki S, Pilcher D, Bellomo R. Mortality related to severe sepsis and septic shock among critically ill patients in Australia and New Zealand, 2000-2012. JAMA. 2014 Apr 2;311(13):1308-16. doi: 10.1001/jama.2014.2637. PMID 24638143
- [Background] Needham DM, Davidson J, Cohen H, Hopkins RO, Weinert C, Wunsch H, Zawistowski C, Bemis-Dougherty A, Berney SC, Bienvenu OJ, Brady SL, Brodsky MB, Denehy L, Elliott D, Flatley C, Harabin AL, Jones C, Louis D, Meltzer W, Muldoon SR, Palmer JB, Perme C, Robinson M, Schmidt DM, Scruth E, Spill GR, Storey CP, Render M, Votto J, Harvey MA. Improving long-term outcomes after discharge from intensive care unit: report from a stakeholders' conference. Crit Care Med. 2012 Feb;40(2):502-9. doi: 10.1097/CCM.0b013e318232da75. PMID 21946660
- [Background] Shao C, Gu L, Mei Y, Li M. [Analysis of the risk factors of cognitive impairment in post-intensive care syndrome patient]. Zhonghua Wei Zhong Bing Ji Jiu Yi Xue. 2017 Aug;29(8):716-720. doi: 10.3760/cma.j.issn.2095-4352.2017.08.009. Chinese. PMID 28795670
- [Background] Pandharipande PP, Girard TD, Jackson JC, Morandi A, Thompson JL, Pun BT, Brummel NE, Hughes CG, Vasilevskis EE, Shintani AK, Moons KG, Geevarghese SK, Canonico A, Hopkins RO, Bernard GR, Dittus RS, Ely EW; BRAIN-ICU Study Investigators. Long-term cognitive impairment after critical illness. N Engl J Med. 2013 Oct 3;369(14):1306-16. doi: 10.1056/NEJMoa1301372. PMID 24088092
- [Background] Jackson JC, Ely EW. Cognitive impairment after critical illness: etiologies, risk factors, and future directions. Semin Respir Crit Care Med. 2013 Apr;34(2):216-22. doi: 10.1055/s-0033-1342984. Epub 2013 May 28. PMID 23716312
- [Background] Jackson JC, Hopkins RO, Miller RR, Gordon SM, Wheeler AP, Ely EW. Acute respiratory distress syndrome, sepsis, and cognitive decline: a review and case study. South Med J. 2009 Nov;102(11):1150-7. doi: 10.1097/SMJ.0b013e3181b6a592. PMID 19864995
- [Background] Trogrlic Z, van der Jagt M, Bakker J, Balas MC, Ely EW, van der Voort PH, Ista E. A systematic review of implementation strategies for assessment, prevention, and management of ICU delirium and their effect on clinical outcomes. Crit Care. 2015 Apr 9;19(1):157. doi: 10.1186/s13054-015-0886-9. PMID 25888230
- [Background] Khan BA, Lasiter S, Boustani MA. CE: critical care recovery center: an innovative collaborative care model for ICU survivors. Am J Nurs. 2015 Mar;115(3):24-31; quiz 34, 46. doi: 10.1097/01.NAJ.0000461807.42226.3e. PMID 25674682
- [Background] Kapfhammer HP, Rothenhausler HB, Krauseneck T, Stoll C, Schelling G. Posttraumatic stress disorder and health-related quality of life in long-term survivors of acute respiratory distress syndrome. Am J Psychiatry. 2004 Jan;161(1):45-52. doi: 10.1176/appi.ajp.161.1.45. PMID 14702249
- [Background] Jackson JC, Pandharipande PP, Girard TD, Brummel NE, Thompson JL, Hughes CG, Pun BT, Vasilevskis EE, Morandi A, Shintani AK, Hopkins RO, Bernard GR, Dittus RS, Ely EW; Bringing to light the Risk Factors And Incidence of Neuropsychological dysfunction in ICU survivors (BRAIN-ICU) study investigators. Depression, post-traumatic stress disorder, and functional disability in survivors of critical illness in the BRAIN-ICU study: a longitudinal cohort study. Lancet Respir Med. 2014 May;2(5):369-79. doi: 10.1016/S2213-2600(14)70051-7. Epub 2014 Apr 7. PMID 24815803
- [Background] Roberts BL, Rickard CM, Rajbhandari D, Reynolds P. Factual memories of ICU: recall at two years post-discharge and comparison with delirium status during ICU admission--a multicentre cohort study. J Clin Nurs. 2007 Sep;16(9):1669-77. doi: 10.1111/j.1365-2702.2006.01588.x. PMID 17727586
- [Background] Garrouste-Orgeas M, Coquet I, Perier A, Timsit JF, Pochard F, Lancrin F, Philippart F, Vesin A, Bruel C, Blel Y, Angeli S, Cousin N, Carlet J, Misset B. Impact of an intensive care unit diary on psychological distress in patients and relatives*. Crit Care Med. 2012 Jul;40(7):2033-40. doi: 10.1097/CCM.0b013e31824e1b43. PMID 22584757
- [Background] Kamdar BB, Huang M, Dinglas VD, Colantuoni E, von Wachter TM, Hopkins RO, Needham DM; National Heart, Lung, and Blood Institute Acute Respiratory Distress Syndrome Network. Joblessness and Lost Earnings after Acute Respiratory Distress Syndrome in a 1-Year National Multicenter Study. Am J Respir Crit Care Med. 2017 Oct 15;196(8):1012-1020. doi: 10.1164/rccm.201611-2327OC. PMID 28448162
- [Background] O'Connor MF, Nunnally ME. Expect the unexpected: clinical trials are key to understanding post-intensive care syndrome. Crit Care. 2013 Jun 12;17(3):149. doi: 10.1186/cc12725. PMID 23759107
- [Background] Pourmand A, Davis S, Lee D, Barber S, Sikka N. Emerging Utility of Virtual Reality as a Multidisciplinary Tool in Clinical Medicine. Games Health J. 2017 Oct;6(5):263-270. doi: 10.1089/g4h.2017.0046. Epub 2017 Jul 31. PMID 28759254
- [Background] Dascal J, Reid M, IsHak WW, Spiegel B, Recacho J, Rosen B, Danovitch I. Virtual Reality and Medical Inpatients: A Systematic Review of Randomized, Controlled Trials. Innov Clin Neurosci. 2017 Feb 1;14(1-2):14-21. eCollection 2017 Jan-Feb. PMID 28386517
- [Background] Larson EB, Ramaiya M, Zollman FS, Pacini S, Hsu N, Patton JL, Dvorkin AY. Tolerance of a virtual reality intervention for attention remediation in persons with severe TBI. Brain Inj. 2011;25(3):274-81. doi: 10.3109/02699052.2010.551648. PMID 21299370
- [Background] Turon M, Fernandez-Gonzalo S, Jodar M, Goma G, Montanya J, Hernando D, Bailon R, de Haro C, Gomez-Simon V, Lopez-Aguilar J, Magrans R, Martinez-Perez M, Oliva JC, Blanch L. Feasibility and safety of virtual-reality-based early neurocognitive stimulation in critically ill patients. Ann Intensive Care. 2017 Dec;7(1):81. doi: 10.1186/s13613-017-0303-4. Epub 2017 Aug 2. PMID 28770543
- [Background] Mosadeghi S, Reid MW, Martinez B, Rosen BT, Spiegel BM. Feasibility of an Immersive Virtual Reality Intervention for Hospitalized Patients: An Observational Cohort Study. JMIR Ment Health. 2016 Jun 27;3(2):e28. doi: 10.2196/mental.5801. PMID 27349654
- [Background] Gerber SM, Jeitziner MM, Wyss P, Chesham A, Urwyler P, Muri RM, Jakob SM, Nef T. Visuo-acoustic stimulation that helps you to relax: A virtual reality setup for patients in the intensive care unit. Sci Rep. 2017 Oct 16;7(1):13228. doi: 10.1038/s41598-017-13153-1. PMID 29038450
- [Background] Sauseng P, Klimesch W, Stadler W, Schabus M, Doppelmayr M, Hanslmayr S, Gruber WR, Birbaumer N. A shift of visual spatial attention is selectively associated with human EEG alpha activity. Eur J Neurosci. 2005 Dec;22(11):2917-26. doi: 10.1111/j.1460-9568.2005.04482.x. PMID 16324126
- [Background] Muller MM, Gruber T, Keil A. Modulation of induced gamma band activity in the human EEG by attention and visual information processing. Int J Psychophysiol. 2000 Dec 1;38(3):283-99. doi: 10.1016/s0167-8760(00)00171-9. PMID 11102668
- [Background] Badcock NA, Mousikou P, Mahajan Y, de Lissa P, Thie J, McArthur G. Validation of the Emotiv EPOC((R)) EEG gaming system for measuring research quality auditory ERPs. PeerJ. 2013 Feb 19;1:e38. doi: 10.7717/peerj.38. Print 2013. PMID 23638374
- [Background] Brummel NE, Jackson JC, Girard TD, Pandharipande PP, Schiro E, Work B, Pun BT, Boehm L, Gill TM, Ely EW. A combined early cognitive and physical rehabilitation program for people who are critically ill: the activity and cognitive therapy in the intensive care unit (ACT-ICU) trial. Phys Ther. 2012 Dec;92(12):1580-92. doi: 10.2522/ptj.20110414. Epub 2012 May 10. PMID 22577067
- [Background] Standen PJ, Threapleton K, Richardson A, Connell L, Brown DJ, Battersby S, Platts F, Burton A. A low cost virtual reality system for home based rehabilitation of the arm following stroke: a randomised controlled feasibility trial. Clin Rehabil. 2017 Mar;31(3):340-350. doi: 10.1177/0269215516640320. Epub 2016 Jul 10. PMID 27029939
- [Background] Saposnik G, Cohen LG, Mamdani M, Pooyania S, Ploughman M, Cheung D, Shaw J, Hall J, Nord P, Dukelow S, Nilanont Y, De Los Rios F, Olmos L, Levin M, Teasell R, Cohen A, Thorpe K, Laupacis A, Bayley M; Stroke Outcomes Research Canada. Efficacy and safety of non-immersive virtual reality exercising in stroke rehabilitation (EVREST): a randomised, multicentre, single-blind, controlled trial. Lancet Neurol. 2016 Sep;15(10):1019-27. doi: 10.1016/S1474-4422(16)30121-1. Epub 2016 Jun 27. PMID 27365261
- [Background] Brown NJ, Rodger S, Ware RS, Kimble RM, Cuttle L. Efficacy of a children's procedural preparation and distraction device on healing in acute burn wound care procedures: study protocol for a randomized controlled trial. Trials. 2012 Dec 12;13:238. doi: 10.1186/1745-6215-13-238. PMID 23234491
- [Background] Salem Y, Elokda A. Use of virtual reality gaming systems for children who are critically ill. J Pediatr Rehabil Med. 2014;7(3):273-6. doi: 10.3233/PRM-140296. PMID 25260510
- See also: Demonstration of the FOVE immersive virtual reality head-mounted display — https://www.youtube.com/watch?v=LNtu5sbrzEA
- See also: Demonstration of the MUSE EEG headband — https://www.youtube.com/watch?v=Ern-WHr4rfI